CLINICAL TRIAL: NCT07096505
Title: The Effects of Early vs. Delayed Time-Restricted Eating on Metabolic Syndrome Parameters in Obese Women: A Randomized Controlled Trial
Brief Title: The Effects of Early vs. Delayed Time-Restricted Eating on Metabolic Syndrome Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SINEM BAYRAM (Other)
Responsible Party: Sponsor-Investigator, SINEM BAYRAM, Assoc. Prof., Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SINEM_TRE_2025; KA23/107 (Other: Başkent University Medical and Health Sciences Research Ethics Committee)
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Obesity and Metabolic Syndrome
Keywords: time restricted eating; obesity; intermittent fasting; randomized controlled trial
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Intermittent Fasting | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A total of 36 obese women aged between 20-49 years were randomly assigned to one of three groups: Early Time-Restricted Eating (eTRE; 08:00-16:00), Delayed Time-Restricted Eating (dTRE; 12:00-20:00), and a Control group (08:00-20:00). A one-day physical activity log was used to assess the participants' physical activity levels. Total energy expenditure was calculated for all participants, and a 25% energy restriction was applied to design individualized medical nutrition therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Time-Restricted Eating with Calorie Restriction (Experimental): Participants ate all meals between 08:00 and 16:00 daily with calorie restriction diet for 8 weeks.
  Interventions: Behavioral: Early time restricted eating with calorie restriction
- Delayed Time-Restricted Eating with Calorie Restriction (Experimental): Participants ate all meals between 12:00 and 20:00 daily with calorie restriction diet for 8 weeks.
  Interventions: Behavioral: Delayed Time Restricted Eating with calorie restriction
- control (Active Comparator): Participants ate all meals between 08:00 and 20:00 daily with calorie restriction diet for 8 weeks.
  Interventions: Behavioral: Control group with calorie restriction

INTERVENTIONS:
Behavioral: Early time restricted eating with calorie restriction — Participants followed a diet with 25% energy restriction and an 8-hour eating window from 08:00 to 16:00. Dietary compliance was monitored by dietitian through food consumption records.
  Arms: Early Time-Restricted Eating with Calorie Restriction
Behavioral: Delayed Time Restricted Eating with calorie restriction — Participants followed a diet with 25% energy restriction and an 8-hour eating window from 12:00 to 20:00. Dietary compliance was monitored by dietitian through food consumption records.
  Arms: Delayed Time-Restricted Eating with Calorie Restriction
Behavioral: Control group with calorie restriction — Participants followed a diet with 25% energy restriction and a usual eating window from 08:00 to 20:00. Dietary compliance was monitored by dietitian through food consumption records.
  Arms: control

SUMMARY:
This study aims to compare the effects of early and delayed time-restricted eating on metabolic syndrome parameters in obese women.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effects of time-restricted eating with different timing windows on metabolic syndrome parameters. A total of 36 sedentary obese women aged between 20-49 years were randomly assigned to one of three groups: Early Time-Restricted Eating (eTRE; 08:00-16:00), Delayed Time-Restricted Eating (dTRE; 12:00-20:00), and a Control group (08:00-20:00). Participants' physical activity levels were assessed using a one-day physical activity log. Total energy expenditure was calculated, and a 25% energy restriction was applied to create individualized medical nutrition therapy. Anthropometric measurements, body composition, and biochemical parameters were collected before and after the 8-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m²
* Able to follow dietary protocols
* No chronic disease (T1DM, T2DM, cardiovascular disease, cancer)
* Not on a weight loss diet in the past 6 months
* No psychiatric disorder
* Sedentary lifestyle

Exclusion Criteria:

* Menopausal women
* Cardiovascular disease
* Type 1 or Type 2 Diabetes
* Use of weight loss medications
* Pregnant or breastfeeding
* Smoking
* Shift workers

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight (kg) | from enrollment to the end of treatment at 8 weeks
  Body weight will be measured in kilograms using standardized procedures at baseline and at the end of the 8-week intervention.
Change in Body Mass Index (BMI) (kg/m²) | from enrollment to the end of treatment at 8 weeks
  Body Mass Index (BMI), calculated as weight (kg) divided by height squared (m²), will be recorded at baseline and at the end of the 8-week intervention.
Change in Waist Circumference (cm) | from enrollment to the end of treatment at 8 weeks
  Waist circumference will be measured in centimeters at baseline and at the end of the 8-week intervention using standardized anthropometric procedures.

SECONDARY OUTCOMES:
Change in Fasting Glucose (mg/dL) | From enrollment to the end of the treatment at 8 weeks
  Fasting blood glucose levels will be measured in mg/dL at baseline and after the 8-week intervention.
Change in Fasting Insulin (μIU/mL) | From enrollment to the end of the treatment at 8 weeks
  Fasting serum insulin levels will be measured in μIU/mL at baseline and after the 8-week intervention.
Change in HOMA-IR | From enrollment to the end of the treatment at 8 weeks
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated using fasting glucose and insulin values at baseline and after the 8-week intervention.
Change in Total Cholesterol (mg/dL) | From enrollment to the end of the treatment at 8 weeks
  Serum Total Cholesterol will be measured in mg/dL at baseline and after the intervention.
Change in Systolic and Diastolic Blood Pressure (mmHg) | From enrollment to the end of the treatment at 8 weeks
  Systolic and diastolic blood pressure will be measured using a standardized sphygmomanometer at baseline and after 8 weeks.
Change in LDL Cholesterol (mg/dL) | From enrollment to the end of the treatment at 8 weeks
  Serum LDL cholesterol will be measured in mg/dL at baseline and after the intervention.
Change in HDL Cholesterol (mg/dL) | From enrollment to the end of the treatment at 8 weeks
  Serum HDL cholesterol will be measured in mg/dL at baseline and after the intervention.
Change in Triglycerides (mg/dL) | From enrollment to the end of the treatment at 8 weeks
  Serum triglyceride levels will be measured in mg/dL at baseline and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Bayram, Assoc. Prof., Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in time-restricted eating and metabolic syndrome. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).